CLINICAL TRIAL: NCT06535256
Title: Comparison of Intraperitoneal Instillation of Bupivacaine with Dexmedetomidine Versus Bupivacaine with Dexamethasone on Postoperative Pain After Laparoscopic Cholecystectomy
Brief Title: Compare Intraperitoneal Instillation of Bupivacaine+dexmedetomidine Versus Bupivacaine+dexamethasone on Postoperative Pain After Lap Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Zaher Zaki Zaher, Lecturer, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Asw 917/5/24
Record Dates: First submitted 2024-07-25; First posted 2024-08-02 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bupivacaine with dexamethasone (Active Comparator): 40 mL of 0.25% bupivacaine + 16 mg dexamethasone with 5 ml normal saline).
  Interventions: Combination Product: bupivacaine with dexamethasone
- bupivacaine with dexmedetomidine (Active Comparator): 40 mL of 0.25% bupivacaine + dexmedetomidine 1 μg/kg with normal saline 5 ml).
  Interventions: Combination Product: bupivacaine with dexmedetomidine

INTERVENTIONS:
Combination Product: bupivacaine with dexamethasone — intra-peritoneal instillation of bupivacaine with dexamethasone (received 40 mL of 0.25% bupivacaine + 16 mg dexamethasone with 5 ml normal saline).
  Arms: bupivacaine with dexamethasone
Combination Product: bupivacaine with dexmedetomidine — intra-peritoneal instillation of bupivacaine with dexmedetomidine (received 40 mL of 0.25% bupivacaine + dexmedetomidine 1 μg/kg with normal saline 5 ml).
  Arms: bupivacaine with dexmedetomidine

SUMMARY:
Comparison of intraperitoneal instillation of bupivacaine with dexmedetomidine versus bupivacaine with dexamethasone on postoperative pain after laparoscopic cholecystectomy

DETAILED DESCRIPTION:
Laparoscopy has become the preferred mode for many diagnostic and operative procedures. It has the advantage better cosmetic results, faster recovery, short post-operative hospital stays, and early resumption of normal activities. Post-laparoscopic pain results from stretching of the intra-abdominal cavity, peritoneal inflammation, and diaphragmatic irritation caused by residual carbon-dioxide in the peritoneal cavity is very annoying to the patients.

Although the severity of pain after a laparoscopic procedure is less compared to laparotomy, but it is acute and can lead to increased analgesic requirements and prolonged hospital stays.

Several studies have evaluated post-laparoscopic pain relief methods such as intravenous analgesics analgesic patches, steroids, and intra-peritoneal instillation of local anaesthetics alone or with additives.

ELIGIBILITY:
Inclusion criteria:

* Patients scheduled for laparoscopic cholecystectomy
* Age 18-60 years
* American Society of Anesthesiologists (ASA) physical status I-II

Exclusion criteria:

* Patients with diabetes mellitus
* Allergy to the study drugs
* Patients on steroids
* Pregnant females
* Patients with cardiac, pulmonary, hepatic or renal disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
incidence and severity of postoperative pain for 24 hours | severity of postoperative pain measured at 1, 2, 4, 8, 16, and 24 hours. postoperatively, using Visual Analogue Scale
  using VAS pain score

CONTACTS AND LOCATIONS:
Locations (1):
- Zaher, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No